CLINICAL TRIAL: NCT05275868
Title: An Open-label, Phase I, Dose Escalation, Expansion Study of MGY825 in Adult Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Study of MGY825 in Patients With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated due to a business decision and not as a result of any safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMGY825A12101; 2023-504350-36-00 (Registry Identifier: CTIS (EU CTR))
Record Dates: First submitted 2022-02-24; First posted 2022-03-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer (NSCLC); NFE2L2; NRF2; KEAP1; CUL3; MGY825
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): Patients with advanced NSCLC harboring NFE2L2/KEAP1/CUL3 mutations enrolled based on locally available test results of mutation status
  Interventions: Drug: MGY825
- Dose expansion group 1 (Experimental): Patients with advanced NSCLC harboring NFE2L2/KEAP1/CUL3 mutations enrolled based on locally available test results of mutation status
  Interventions: Drug: MGY825
- Dose expansion group 2 (Experimental): Patients with advanced NSCLC irrespective of prior knowledge of NFE2L2/KEAP1/CUL3 mutational status.
  Interventions: Drug: MGY825

INTERVENTIONS:
Drug: MGY825 — investigational drug

SUMMARY:
Study of MGY825 single agent in adult patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
First in human, phase I, multicenter, open-label study of MGY825 single agent with a dose escalation and a dose expansion in adult patients with advanced non-small cell lung cancer (NSCLC).

The dose escalation part investigated the safety and tolerability of MGY825 in adult patients with advanced NSCLC harboring NFE2L2, or KEAP1 or CUL3 (NFE2L2/KEAP1/CUL3) mutations. Patient enrollment was based on locally available test results of mutation status.

An exploratory assessment on the effect of food could be investigated during the dose escalation part.

The dose expansion part assessed the preliminary anti-tumor activity and further assess the safety and tolerability of MGY825 in adult patients with advanced NSCLC divided in two patient groups.

Group 1: Patients with advanced NSCLC harboring NFE2L2/KEAP1/CUL3 mutations enrolled based on locally available test results of mutation status.

Group 2: Patients with advanced NSCLC irrespective of prior knowledge of NFE2L2/KEAP1/CUL3 mutational status.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Dose escalation and dose expansion group 1:

Patients with histologically or cytologically confirmed diagnosis of advanced (metastatic or unresectable) NFE2L2/KEAP1/CUL3 mutant NSCLC. Local data confirming the NFE2L2/KEAP1/CUL3 mutation status in tissue must be available for enrollment.

* Dose expansion group 2:

Patients with histologically or cytologically confirmed diagnosis of advanced (metastatic or unresectable) NSCLC irrespective of NFE2L2/KEAP1/CUL3 mutation status.

* All patients:

Patients must have progressed after 1 platinum-based chemotherapy regimen and PD-(L)1 antibody therapy either sequentially or concurrent with chemotherapy, where indicated, for Stage IV NSCLC.

Patients treated with neo-adjuvant / adjuvant platinum-based therapy that progressed within 6 months of treatment are permitted to participate.

Prior therapy with VEGF/VEGFR targeting agents is permitted. Prior treatment with approved targeted drugs (e.g., EGFRi, ALKi, METi) is mandatory in patients with NSCLC whose tumor bears actionable mutations.

* Presence of at least one measurable lesion according to RECIST v1.1.
* Patient must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening and during study treatment. A recent biopsy collected after the last systemic treatment and within 3 months before study entry may be submitted at screening.

Exclusion Criteria:

* Having out of range laboratory values defined as:

Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 60 mL/min Total bilirubin > 1.5 x ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN ALT > 3 x ULN AST > 3 x ULN ANC < 1.0 x 109/L Platelet count < 75 x 109/L Hemoglobin < 9 g/dL

* Impaired cardiac function or clinically significant cardiac disease, including any of the following:

Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥2), uncontrolled hypertension or clinically significant arrhythmia.

QTcF > 470 msec on screening ECG or congenital long QT syndrome. Acute myocardial infarction or unstable angina pectoris < 3 months prior to study entry.

* Presence of symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery) or increasing doses of corticosteroids within 2 weeks prior to study entry. Patients with treated symptomatic brain metastases should be neurologically stable (for 4 weeks post-treatment and prior to study entry) and at a dose of ≤ 10 mg per day prednisone or equivalent for at least 2 weeks before administration of any study treatment.
* Known active COVID-19 infection.
* Unable or unwilling to swallow capsules as per dosing schedule. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 28 months
  Assessment of safety of study drug as a single agent
Frequency of dose interruptions and reductions | 28 months
  Assessment of tolerability of study drug as a single agent
Dose intensity | 28 months
  Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of exposure.
Incidence and nature of dose limiting toxicities (DLTs) during the first 28 days of treatment with the study drug | 28 days
  A DLT is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 assessed as not primarily related to disease, disease progression, inter-current illness or concomitant medications that occurs during the first 28 days of treatment with the study drug. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | 20 months
  Pharmacokinetics (PK) parameters will be determined by non-compartmental methods using the PK profile of the study drug.
Peak concentration (Cmax) | 20 months
  Pharmacokinetics (PK) parameters will be determined by non-compartmental methods using the PK profile of the study drug.
Time to reach maximum drug concentrations in systemic circulation (Tmax) | 20 months
  Pharmacokinetics (PK) parameters will be determined by non-compartmental methods using the PK profile of the study drug.
Overall response rate (ORR) per RECIST 1.1 | 28 months
  Evaluation of preliminary anti-tumor activity of study drug as single agent
Progression free survival (PFS) per RECIST 1.1 | 28 months
  Evaluation of preliminary anti-tumor activity of study drug as single agent
Duration of response (DOR) per RECIST 1.1 | 28 months
  Evaluation of preliminary anti-tumor activity of study drug as single agent

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wash U School of Medicine, St Louis, Missouri
  - NYU School of Medicine, New York, New York
  - Memorial Sloan Kettering Onc. Dept, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Germany (3):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Madrid, Spain
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No